CLINICAL TRIAL: NCT01979510
Title: A Phase III Randomized Clinical Trial to Evaluate the Safety and Efficacy of an Etoricoxib and Tizanidine Fixed Dose Combination in Subjects With Moderate to Severe Acute Low Back Pain
Brief Title: Safety and Efficacy Study of an Etoricoxib and Tizanidine Fixed Dose Combination in Participants With Moderate to Severe Acute Low Back Pain (MK-0663B-164)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663B-164
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MK-0663B (Experimental): MK-0663B (etoricoxib 90 mg immediate release [IR]/tizanidine 6 mg modified release [MR]) capsules once daily for 8 days.
  Interventions: Drug: MK-0663B; Drug: Acetaminophen 500 mg
- DOLOCAM PLUS® (Experimental): DOLOCAM PLUS® (meloxicam 7.5mg/methocarbamol 215mg) capsules once daily for 8 days.
  Interventions: Drug: DOLOCAM PLUS®; Drug: Acetaminophen 500 mg

INTERVENTIONS:
Drug: MK-0663B — MK-0663B once daily for 8 days.
  Arms: MK-0663B
Drug: DOLOCAM PLUS® — DOLOCAM PLUS® once daily for 8 days.
  Arms: DOLOCAM PLUS®
Drug: Acetaminophen 500 mg — Acetaminophen 500 mg up to 4 times daily for up to 8 days as required for uncontrolled breakthrough pain.

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of MK-0663B (etoricoxib/tizanidine) among participants with moderate-to-severe acute low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Have acute low back pain;
* Onset of acute low back pain must be <6 weeks prior to screening;
* Have acute low back pain corresponding to a rating of ≥ 4 on a 0-10 point Low Back Pain Questionnaire and ≥ 7 on the Roland Morris Questionnaire;
* For women of childbearing potential, have a negative serum pregnancy test at Visit 1 (Screening Visit) and agree to remain abstinent, use barrier, or non-hormonal implanted contraceptives from study start until 14 days after the last dose of study drug;
* Be willing to limit alcohol use, if any, to 2 drinks or equivalent per day for the duration of the study and follow-up period;
* Be willing to avoid unaccustomed physical activity (e.g., starting a new weight lifting routine) for the duration of the study and follow-up period;
* Be willing to avoid chiropractic care, ultrasound and physical therapy from screening to Day 9;
* Be willing to avoid cold applications and other alternate treatments (e.g. massage, acupuncture etc.) on Day 1 and within 30 minutes prior to scheduled pain assessments on Day 3 and Day 8.

Exclusion Criteria:

* Has low back pain that is related to, or known to be caused by malignancy, inflammatory disease (rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, Reiter's syndrome), osteoporosis, ochronosis, vertebral fracture, infection, juvenile scoliosis, congenital malformation, or fibromyalgia. Note: the presence of radiographic degenerative disc disease is not an exclusion;
* Has signs or symptoms consistent with a neurologic, infectious, or fracture-related cause of acute low back pain;
* Has chronic low back pain and is experiencing an acute flare-up of the chronic back pain condition;
* Has radicular or myelopathic pain;
* Has a history of lumbar spine surgery;
* Is involved in an active civil lawsuit or workman's compensation claim pertaining to his/her low back pain;
* Has symptomatic depression that could interfere with the completion of the questionnaires;
* Is mentally or legally incapacitated, has significant emotional problems at the time of the study, or has a history of major psychiatric disorder, including any history of psychosis;
* Has a Body Mass Index (BMI) ≥ 40;
* Is allergic to, or has a history of a significant clinical or laboratory adverse experience associated with tizanidine, etoricoxib, methocarbamol, meloxicam, or any non-steroidal anti-inflammatory drug (NSAID);
* Is allergic to acetaminophen/paracetamol;
* Is currently a user (including "recreational use") of any illicit drugs, or has a history (within 5 years) of drug or alcohol abuse;
* Has participated in another investigational drug study within the last 4 weeks;
* Has uncontrolled hypertension;
* Has systolic blood pressure (SBP) < 105 or diastolic blood pressure (DBP) < 65;
* Has a history of orthostatic hypotension;
* Has ischemic heart disease, peripheral arterial disease and/or cerebrovascular disease;
* Has a positive human immunodeficiency virus (HIV) test result, hepatitis B surface (HBS) antigen, or hepatitis C virus (HCV) test result;
* Has a history of hepatitis/hepatic disease that has been active within the previous year;
* Has a history of gastric, biliary, or small intestinal surgery or disease that results in clinical malabsorption;
* Has a history of neoplastic disease;
* Has any personal or family history of an inherited or acquired bleeding disorder;
* Is expected to undergo a planned surgical procedure or invasive diagnostic procedure during the course of the study;
* Is pregnant or breast-feeding, or expecting to conceive within the projected duration of the study;
* Has an active peptic ulcer or a history of inflammatory bowel disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing an Adverse Event (AE) | Up to Day 23
Number of Participants Discontinuing Study Treatment Due to an AE | Up to Day 8

SECONDARY OUTCOMES:
Mean Change From Baseline in the Participant Low Back Pain Questionnaire Score | Baseline and Day 9
Mean Change From Baseline in the Participant Roland Morris Disability Questionnaire | Baseline and Day 9
Number of Participants With ≥30% Improvement From Baseline in the Roland Morris Disability | Baseline and Day 9
Mean Change From Baseline in the Participant Global Assessment of Response to Therapy. | Baseline and Day 9
Mean Change From Baseline in the Investigator Global Assessment of Response to Therapy | Baseline and Day 9
Average Amount of Rescue Medication Required by Participant During Study Treatment | Up to Day 8
Proportion of Participants Using Rescue Medication During Study Treatment | Up to Day 8